CLINICAL TRIAL: NCT02232009
Title: Development of MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit
Brief Title: Development of a MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit
Acronym: Firefly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow/low enrollment
Sponsor: GE Healthcare (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114-2013-GES-0011
Record Dates: First submitted 2014-08-15; First posted 2014-09-04 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Image Evaluation
Keywords: Neonate; Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3.0 T Neonatal Scanner (Other): All subjects who participate in this study will be scanned using the 3.0 T Neonatal MRI scanner.
  Interventions: Device: 3.0 T Neonatal MRI Scanner

INTERVENTIONS:
Device: 3.0 T Neonatal MRI Scanner — Eligible subjects will undergo neonatal MRI scanning procedures.

SUMMARY:
This study investigates a novel magnetic resonance imaging (MRI) system designed by GEHC for imaging viable neonate and infant populations. This MR system has a smaller size and design features that may make it more feasible to locate the system in close proximity to care areas for neonates (birth - 1 month) and infants (less than 1 month to two years), such as clinical neonatal intensive care units (NICUs) and other infant and neonatal care departments.

DETAILED DESCRIPTION:
This study investigates a novel magnetic resonance imaging (MRI) system designed by GEHC for imaging viable neonate and infant populations. This MR system has a smaller size and design features that may make it more feasible to locate the system in close proximity to care areas for neonates (birth - 1 month) and infants (>1 month to two years), such as clinical neonatal intensive care units (NICUs) and other infant and neonatal care departments.

This is a two-phase prospective clinical study evaluating the performance and safety of the investigational MRI device for neonates and infants, including:

* Phase 1 - Initial feasibility assessment and optimization study (Phase 1) which may include hardware and software modifications. These studies are guided by a series of MR scanning procedures defined in sequential Sponsor-provided MR Procedure Documents
* Phase 2 - Controlled image and data collection study based on Phase 1 results, in which optimized scan procedure(s) according to MR Procedure Document(s) will be provided at the start of Phase 2 scanning and a fixed hardware and integrated software configuration will be applied for all subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included that are:

1. Currently admitted for treatment or observation at the investigational site at the time of enrollment;
2. In the weight range less than 5.0 kg (<5.0 kg ) and more than 0.5 kg (>0.5 kg );
3. Viable neonates (birth to 1 month of age) or infants (>1 month to two years of age);
4. Able to safely undergo an MRI scan, as determined by the site's co-investigator neonatologist or medically qualified delegate;
5. Have parent(s), guardian(s), or legally authorized representative(s) willing and able to provide written informed consent for the subject's participation;
6. Are of appropriate size and shape to fit into the bore of the magnet, inclusive of all monitoring equipment, if any, necessary for the subject's routine clinical care:

   1. Maximum width (shoulder-to-shoulder measurement) less than eighteen (18 cm).
   2. Maximum length (head-to-foot measurement) less than sixty (60) cm. -

Exclusion Criteria:

* Subjects will be excluded that:

  1. Have parent(s), guardian(s), or legally authorized representative(s) that require that they accompany the subject into the MR environment that have contraindications to the MR environment or would otherwise be put at undue risk or discomfort, as determined by the investigators;
  2. Require any non-removable medical devices that are not compatible with MR scanning (labeled as MR Unsafe, MR condition for which the scanning conditions are not met, or no MR safety labeling) that may pose hazards in the MR scanning or MR environment, in the opinion of the neonatologist co-investigator or medically qualified delegate;
  3. Have other contraindications or could otherwise be expected to experience detrimental effects to safety, well-being, or medical care, as determined by the neonatologist co-investigator;
  4. Require any scheduled standard of care procedures that are expected to be adversely impacted by participation in this study, in the opinion of the principal investigator, neonatologist co-investigator, or medically qualified delegate; and
  5. Have been previously enrolled AND undergone any study procedures under the current study protocol (i.e. the same subject cannot undergo study procedures, including swaddling and/or MR scanning, more than once).

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3.0 T Neonatal Scanner
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Summary Rates of Adverse Events
Description: Safety will be assessed based on the number of Adverse Events.
Time Frame: 1 Day
Measure: Number; unit: number of occurrences
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
number of occurrences | 1

2. Primary Outcome: Image Diagnostic Quality
Description: Number of subject whose images were rated as Evaluable
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: MRI Scan Time
Description: Duration of MRI scan time for each subject
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
minutes | 57 (6.08)

4. Secondary Outcome: Overall Experience With Neonatal MR Scanner Device Summary
Description: User survey results on a scale from 1 to 5, where 1 = strongly disagree and 5 = strongly agree.
Time Frame: 1 day
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
score on a scale
  Like to use frequently | 3.22 [1 to 4]
  Unnecessarily complex | 3.11 [2 to 4]
  Easy to Use | 2.56 [2 to 4]
  Would need tech support to use | 3.00 [2 to 4]
  Functions are well integrated | 2.89 [2 to 4]
  Too much inconsistency | 2.78 [2 to 4]
  Most people would learn quickly | 3.00 [2 to 4]
  Cumbersome to use | 3.0 [2 to 4]
  Felt confident using | 3.0 [2 to 4]
  Needed to learn a lot before using | 3.22 [2 to 4]
  System meets patients needs | 3.56 [3 to 4]
  Would recommend to others | 3.44 [2 to 4]

5. Secondary Outcome: Overall Image Quality
Description: Scores range from 1-Very Poor image quality to 5-Excellent image quality.
Time Frame: 1 day
Measure: Number; unit: Frequency of ratings
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
Frequency of ratings
  1-Very Poor | 0
  2-Poor | 0
  3-Neutral | 3
  4-Good | 6
  5-Excellent | 0

6. Secondary Outcome: Subject Change in Temperature
Description: Change in temperature (Celsius) per subject.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | 3.0 T Neonatal Scanner
Number analyzed (Participants) | 9
Degrees Celsius | -0.07 (0.23)

ADVERSE EVENTS:
Arm/Group | 3.0 T Neonatal Scanner
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.0 T Neonatal Scanner (N=9)
Redness behind ears (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No